CLINICAL TRIAL: NCT00930709
Title: Botulinum Toxin Versus Active Strength Training in Treatment of the Lateral Epicondylitis - A Single-Blinded, Randomized, Controlled Trial
Brief Title: Botulinum Toxin Versus Active Strength Training in the Treatment of Lateral Epicondylitis
Acronym: BooST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Aki Vainionpaa, Specialist in Physical Medicine and Rehabilitation, Seinajoki Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVO1122; 2009-009837-14 (EudraCT Number)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Epicondylitis, Lateral Humeral; Tennis Elbow
Keywords: Botulinum Toxin Type A; Exercise; Randomized Controlled Trial; Muscle Stretching Exercises; Strength Training; Treatment Outcome
MeSH Terms: conditions — Tennis Elbow; Motor Activity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active strength training and stretching (Active Comparator): Active strength training and stretching
  Interventions: Behavioral: Active strength training and stretching
- Botulinum toxin type A injections (Active Comparator): Botulinum toxin type A injections
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan)

INTERVENTIONS:
Drug: Botulinum toxin type A (Botox®, Allergan) — Two injections of 10-60 units of botulinum toxin type A. Injections are administered with ENMG assisted technique at the baseline and after 13 weeks.
  Other Names: Botox®, Allergan; NDC 0023-1145-01
  Arms: Botulinum toxin type A injections
Behavioral: Active strength training and stretching — Training duration 9 weeks, intensified every 3 weeks in supervision of physiotherapist. Training program includes progressive, slow, repetitive wrist and forearm stretching, eccentric muscle strengthening, occupational exercises and upper limb neural mobilization training.
  Other Names: Eccentric strength training
  Arms: Active strength training and stretching

SUMMARY:
The purpose of this study is to compare efficacy, feasibility and cost effectiveness of botulinum toxin type A injections to active nine weeks strength training and stretching program in the treatment of the chronic lateral epicondylitis.

The main hypothesis is that the botulinum toxin type A injections may enable more rapid pain relief while strength training may provide better functional results and less relapses during the follow-up.

DETAILED DESCRIPTION:
INTRODUCTION:

Lateral epicondylitis (tennis elbow) is a frequent repetitive stress injury, affecting the common extensor muscles at the lateral humeral epicondyle. Lateral epicondylitis has a well-known spontaneous healing tendency. Still the prevalence of the chronic lateral epicondylitis is 1.4% in working populations causing significant occupational disability and financial burden.

Systematic reviews of the effectiveness of different treatment modalities for lateral epicondylitis present conflicting results. There are no consistent guidelines for management of the prolonged lateral epicondylitis. Progressive strengthening and stretching exercises as well as botulinum toxin type A injections have been suggested to be effective in treatment of chronic cases. However, there are only a few studies comparing different treatment modalities and botulinum toxin treatment have not been included in any of these.

The purpose of this study is to compare efficacy, feasibility and cost effectiveness of the botulinum toxin type A injections to active nine weeks strength training and stretching program in the treatment of the chronic lateral epicondylitis.

The main hypothesis is that the botulinum toxin type A injections may enable more rapid pain relief while strength training may provide better functional results and less relapses during the follow-up.

SUBJECTS AND METHODS:

A sample size of 120 participants with an equal drop-out rate of 15 % per group was determined in advance to detect a clinically significant 30 percentage points difference in outcome measures between the treatment groups with the minimum success rate of 65 % at the statistical significance level of 0.05 and power of 80 %.

During the recruitment process all patient newly referred to Department of PM&R outpatient clinics in the Seinäjoki Central Hospital due to elbow pain are evaluated by the study investigators. Every eligible patient with written informed consent is recruited. A computerised random number generator is used to draw up an allocation schedule. Patients are allocated in treatment groups via opaque sealed envelopes marked according to the random schedule.

Measurements and training instructions are performed by five trained physical therapists. In addition to detailed personal training instructions given by physical therapist, illustrated instructions as well as instruction video will be provided for patients in the training group. Physical therapists instructing patients do not perform any measurements to enable blinding of assessor. Measurement devices are calibrated regularly according to the manufacturers' recommendations and quality assurance measurements with test weights are performed on regular basis.

The principal statistical analysis will be done on an intention-to-treat basis. Repeated measures of ANCOVA and Cox Proportional Hazard Regression are planned to be used as primary methods. If there will be relapses, more advanced longitudinal models such as Generalised Estimating Equations and Random Coefficient Analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* pain at the lateral side of the elbow over 3 months
* local tenderness on palpation over the lateral epicondyle
* positive Mill's sign
* lateral elbow pain progression on resisted wrist and/or middle finger extension
* involved in working life

Exclusion Criteria:

* bilateral symptoms or simultaneous medial epicondylitis
* verified or suspected cervical radiculopathy or affected limb neuropathy
* congenital or acquired deformities of the elbow
* previous surgery of the elbow
* infection, dislocation, tendon ruptures, or fractures in the area
* systemic musculoskeletal or neurological disorders, incl. rheumatic diseases and fibromyalgia
* allergy, antibodies or other contraindications for botulinum toxin
* severe depression, chronic pain syndrome or somatisation disorder
* ongoing retirement process
* pregnancy or breastfeeding
* current participation in other clinical trials

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain, 100 mm visual analogue scale, change from baseline | 0, 6, 13, 26, 39, 52 weeks
Grip strength (pain free and maximal), hydraulic hand dynamometer, change from baseline | 0, 6, 13, 26, 39, 52 weeks

SECONDARY OUTCOMES:
Experienced disability, 100 mm visual analogue scale, change from baseline | 0, 6, 13, 26, 39, 52 weeks
Isometric wrist extension and flexion strength, digital hanging scale with rigid bench frame, change from baseline | 0, 6, 13, 26, 39, 52 weeks
Treatment adverse effects | 0, 6, 13, 26, 39, 52 weeks
Economic evaluation of interventions, direct and indirect costs | 0, 6, 13, 26, 39, 52 weeks
Days in sick leave | 0, 6, 13, 26, 39, 52 weeks
Experienced forearm pain and disability, The Patient-Rated Tennis Elbow Evaluation (PRTEE) | 0, 6, 13, 26, 39, 52 weeks
General improvement, 7-point Likert scale | 0, 6, 13, 26, 39, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aki Vainionpää, M.D., Ph.D., Principal Investigator — Department of Physical Medicine and Rehabilitation, Seinäjoki Central Hospital
Locations (1):
- Department of Physical medicine and Rehabilitation, Seinäjoki Central Hospital, Seinäjoki, Finland

REFERENCES:
- See also: Seinäjoki Central Hospital homepage — http://www.epshp.fi/